CLINICAL TRIAL: NCT06427434
Title: Effect of Modified Lumbar Sustained Natural Apophyseal Glide on Low Back Pain in Postnatal Women
Brief Title: Effect of Modified Lumbar Sustained Natural Apophyseal Glide on Postnatal Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Nageib Soliman, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004494
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening and stretching exercises (Active Comparator): The participants will be asked to perform strengthening and stretching exercises to the back and abdominal muscles for 30 min, three times per week for 4 weeks.
  Interventions: Other: Strengthening and stretching exercises to the back and abdominal muscles
- Modified Lumbar Sustained Natural Apophyseal Glide (Experimental): The participants will receive Modified Sustained Natural Apophyseal Glide on the affected lumbar level for 30 sec three times per week for 4 weeks. In addition to strengthening and stretching exercises to the back and abdominal muscles for 30 min, three times per week for 4 weeks
  Interventions: Other: Strengthening and stretching exercises to the back and abdominal muscles; Other: Modified Lumbar Sustained Natural Apophyseal Glide

INTERVENTIONS:
Other: Strengthening and stretching exercises to the back and abdominal muscles — Strengthening and stretching exercises to the back and abdominal muscles will be performed for 30 min, three times per week for 4 weeks.
Other: Modified Lumbar Sustained Natural Apophyseal Glide — Modified Sustained Natural Apophyseal Glide will be applied on the affected lumbar level for 30 sec three times per week for 4 weeks.
  Arms: Modified Lumbar Sustained Natural Apophyseal Glide

SUMMARY:
This study will be carried out to evaluate the effect of modified lumbar Sustained Natural Apophyseal Glide on low back pain in postnatal women.

DETAILED DESCRIPTION:
In fact, up to 75% of women who suffer from pregnancy-related back pain may continue to have pain after giving birth. Women who experience LBP or pelvic girdle pain (PGP) at 3 months postpartum were found to be at higher risk for persistent or chronic LBP. Of these women, only 6% recover within 6-18 months after giving birth.

A modified lumbar Sustained Natural Apophyseal Glide (SNAG) is an existing Mulligan mobilization technique performed with a combination of joint glide and physiological spinal movement. The glide can be applied to the spinous processes, facets, or unilaterally over the transverse processes while the patient performs the active exercise.

Few studies have been concerned with the effects of modified "SNAGS" on the lumbar spine . So, this study will be done to investigate its effect on low back pain in postnatal women aiming to improve their function to accomplish their daily living activities and reduce the side effects of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be diagnosed as chronic postnatal low back pain.
2. Their ages will be ranged from 20 to 35 years old.
3. Their body mass index (BMI) will not exceed 30 kg/m2.
4. All participants have the same social level.
5. All participants have the same lifestyle.
6. Their number of parity will be ranged from 2-4 children.

Exclusion Criteria:

1. Spinal fracture or any other neurological disorders.
2. Lumbar spinal stenosis from lumbar disc herniation, degenerative joint diseases, or spondylolisthesis.
3. Women with BMI > 30 kg/m2.
4. Participants who had pelvic pathology.
5. Skin disease interferes with mobilization application.
6. Gynecological diseases (chronic pelvic pain, uterine prolapse and retroversion flexion of the uterus).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pain intenesity | within 4 weeks
  The visual analogue scale is a 10 cm calibrated line with 0 representing no pain and 10 representing the worst pain; will be used to assess the severity of pain before and after treatment for all participants in both groups.
Lumbar flexion range of motion | within 4 weeks
  The modified Schober test will be used to measure the lumbar flexion range of motion (ROM) by using the tape measurement. Each participant will be asked to stand erect with her feet about shoulder-width apart to stabilize the pelvis. Then, the posterior superior iliac spines(PSIS) will be determined by the therapist's both thumbs, and then an ink line will be drawn along the midline of the lumbar spines horizontal to the PSIS to mark the midpoint between the two PSIS. Then tape will be used to identify and mark two points: one is 10 cm superior to the midpoint (A), and another is 5 cm inferior to the midpoint (B). The participant will be instructed to bend forward as much as she can while keeping both knees straight, the new distance between superior and inferior skin marking will be measured in centimeters. The increased distance along the tape due to lumbar flexion is normally about 6-7 cm (less than 5 cm should be considered abnormal).
Lumbar extension range of motion | within 4 weeks
  The modified Schober test will be used to measure the lumbar extension range of motion (ROM) by using the tape measurement while the patient is in a standing position.
  The participant will be instructed to put her hands on her buttocks and bend backward into full lumbar extension and the new distance between the superior and inferior skin markings will be measured in centimeters by the tape measurement. The change in the difference between the marks is used to indicate the amount of lumbar extension.
  The increased distance along the tape due to the extension of the lumbar spine is normally about 2-3 cm (less than 1 cm should be considered abnormal).
Lumbar lateral flexion range of motion | within 4 weeks
  The participant will be asked to stand erect with her feet about shoulder-width apart. Both right and left lateral flexion will be measured by the tape as the distance from the tip of the index finger to the floor at maximal comfortable lateral flexion. The participant will be instructed to bend her trunk laterally as much as she can. The normal value of lateral spinal flexion is 16.2-28.0 cm.

SECONDARY OUTCOMES:
Functional disability | within 4 weeks
  Functional disability will be assessed by the Oswestry Disability Index, it was developed as a clinical valid and reliable assessment tool that would provide an estimate of disability expressed as a percentage score. It is composed of 10 questions and it takes around 5min for a patient to complete. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, bed-bound. A low score = low degree of disability, a high score = high degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Kassab, professor, Study Director — Cairo University
Locations (1):
- Mina Nageb Soliman, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol